CLINICAL TRIAL: NCT00134485
Title: Phase 3, Multi-Center, Double-Blind, Randomized, Parallel Group, Study of the Efficacy, Safety, and Tolerability of Fixed Combination Torcetrapib (CP-529,414) / Atorvastatin Administered Orally, Once Daily (QD) for Six Months, Compared With Maximally Tolerated Atorvastatin Therapy Alone, in Subjects With Heterozygous Familial Hypercholesterolemia
Brief Title: Study To Evaluate The Safety And Efficacy Of Torcetrapib/Atorvastatin In Subjects With Familial Hypercholerolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A5091026
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2007-10-30 (Estimated); Status verified 2006-12

CONDITIONS: Hypercholesterolemia, Familial; Hyperlipidemia
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hyperlipidemias | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: torcetrapib/atorvastatin
Drug: atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To evaluate the efficacy and safety of torcetrapib/atorvastatin compared to atorvastatin alone in patients with heterozygous familial hypercholesterolemia

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Heterozygous Familial Hypercholesterolemia
* At least 18 years of age

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid (high doses)
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluation of response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400
Dates: Start 2005-03; Study Completion 2006-03

PRIMARY OUTCOMES:
Change in HDL-C and LDL-C

SECONDARY OUTCOMES:
Changes in other lipid parameters

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (39):
- United States (14):
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Lutz, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Tripler AMC, Hawaii
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Auburn, Maine
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Madison, Wisconsin
- Australia (6):
  - Pfizer Investigational Site, Camperdown, New South Wales
  - Pfizer Investigational Site, Woolloongabba, Queensland
  - Pfizer Investigational Site, North Adelaide, South Australia
  - Pfizer Investigational Site, Clayton, Victoria
  - Pfizer Investigational Site, Perth, Western Australia
  - Pfizer Investigational Site, Darlinghurst
- Canada (3):
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Montreal, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec
- Denmark (2):
  - Pfizer Investigational Site, Aalborg
  - Pfizer Investigational Site, Arhus C
- France (3):
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Paris
- Pfizer Investigational Site, Kopavogur, Iceland
- Pfizer Investigational Site, Oslo, Norway
- South Africa (4):
  - Pfizer Investigational Site, Parow, Cape Town
  - Pfizer Investigational Site, Bellville, Western Cape
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town
- Sweden (4):
  - Pfizer Investigational Site, Gothenburg
  - Pfizer Investigational Site, Linköping
  - Pfizer Investigational Site, Malmo
  - Pfizer Investigational Site, Stockholm
- Pfizer Investigational Site